CLINICAL TRIAL: NCT06261476
Title: Safety of Ashwagandha (Withania Somnifera) Root Extract: An Open-Label, Non-Comparative, Prospective Study in Healthy Subjects
Brief Title: Safety of Ashwagandha (Withania Somnifera) Root Extract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DYP-Pharm-RP-23
Record Dates: First submitted 2024-01-24; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Ashwagandha

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ashwagandha (Withania somnifera) Root Extract (Experimental): Participants will take two Ashwagandha capsules containing 500 mg standardized root extract twice daily after breakfast and dinner, for a duration of 12 weeks.
  Interventions: Dietary Supplement: Ashwagandha (Withnia somnifera)

INTERVENTIONS:
Dietary Supplement: Ashwagandha (Withnia somnifera) — Ashwagandha is the active ingredient in Withania somnifera (a medicinal plant in Indian medicine). Ashwagandha is known as an adaptogen, an herb in capsule form that protects the body from stress.

SUMMARY:
The primary objective is to evaluate the laboratory safety of Ashwagandha standardized root extract 500 mg capsules in healthy adults over 12-week therapy based on Complete Blood Count, Renal Function Test, Liver Function Test, Lipid Profile and Thyroid Function Test, Fasting blood sugar and HbA1c Test. The secondary objectives are to evaluate the clinical safety of Ashwagandha standardized root extract 500 mg capsules in healthy adults over 12-week therapy and to evaluate the effect of the Ashwagandha standardized root extract 500 mg on Quality of Life (QoL) using the SF-36 tool.

DETAILED DESCRIPTION:
To qualify for this study, participant must be a healthy male or female between 18 and 65 years old, free from any chronic illness, such as diabetic, cardiovascular, or any other conditions that could affect the safety of the study. Participants must have no plan to commence any other alternative treatment modality for their conditions. Participants must be willing to sign an informed consent document and to comply with all study related procedures.

In this study, 100 subjects will be enrolled at 2 sites, for a total duration of 12 weeks. At the initial visit, prospective patients will be screened for enrollment based on the requirements of the study, medical history, and clinical examination. Before starting any study related procedures, participants will be explained about the study in detail and a written informed consent will be obtained from participants prior to participation in this study. This document is a part of the written informed consent procedure. A detailed medical history including the associated conditions will be recorded. A general and physical examination will be performed to detect any abnormal parameters. If participants meet the eligibility criteria, they will be enrolled in the study.

After enrollment in the study, participants will be assigned to take two capsules of Ashwagandha (500 mg) twice daily after breakfast and dinner with ambient temperature water for 12 weeks. At Visit 1 (Screening/Enrollment/Baseline Visit - Day -3 to Day 0), demography and medical history will be taken, physical examination and vital signs will be performed, blood will be collected, and the study medication will be dispensed.

At Visit 2 (Week 4 ± 4 days) and Visit 3 (Week 8 ± 4 days), participants will return to the site for a followup. A physical examination and vital signs will be performed, blood will be collected, study medication will be dispensed, and compliance will be assessed.

At Visit 4 (Final Visit - Week 12 ± 4 days), physical examination and vital signs will be performed, blood will be collected, Quality of Life will be assessed using the SF-36 QoL scale, and compliance will be assessed. Participants will be monitored throughout the study, including any adverse events. At study completion, participants are required to return any remaining testing products to the San Francisco Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Both adults (male and female) aged between 18 and 65 years.
* Participant should be healthy and free from any chronic illness, such as diabetic, cardiovascular or any other condition that could affect the safety of the study.
* No plan to commence any other alternative treatment modality for their conditions.
* Willingness to sign an informed consent document and to comply with all study related procedures.

Exclusion Criteria:

* History of Alcohol or smoking abuse.
* History of hypersensitivity to Ashwagandha.
* Taking nutritional or energy supplements, medication, or steroids.
* Any history of drug abuse.
* Having any clinical abnormalities.
* Simultaneously participating in any other clinical trial or participated in the past three months.
* Participants who use medication for blood pressure, use betablockers, inhaled any beta-agonists, use any hormonal contraceptives, having a history of corticosteroid use within three months, participants under psychotropic medication within last 8 weeks, and
* Participants diagnosed with any heart disease, diabetes, stroke, neurological disorders or depression.
* Have clinically significant acute unstable hepatic, renal, cardiovascular, or respiratory disease that will prevent participation in the study.
* Patients with depressive episode, panic disorder, social phobia, obsessive-compulsory disorder, alcohol dependency; schizophrenia and mania.
* Patients with post traumatic disorder.
* Have an established practice of meditation for three or more months.
* Pregnant and lactating women.
* Participation in other clinical trials during previous 3 months.
* Any clinical condition, according to the investigator which does not allow safe fulfillment of clinical trial protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin Test | 12 weeks
  Evaluate the mean change in hemoglobin from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Total Erythrocyte Count | 12 weeks
  Evaluate the mean change in total erythrocytes from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Total Leukocyte Count | 12 weeks
  Evaluate the mean change in total leukocytes from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Platelet Count | 12 weeks
  Evaluate the mean change in platelets from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Hematocrit Test | 12 weeks
  Evaluate the mean change in hematocrit from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Total Cholesterol Test | 12 weeks
  Evaluate the mean change in total cholesterol from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
LDL Test | 12 weeks
  Evaluate the mean change in LDL from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
HDL Test | 12 weeks
  Evaluate the mean change in HDL from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Triglycerides Test | 12 weeks
  Evaluate the mean change in triglycerides from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Serum Alkaline Transaminase Test | 12 weeks
  Evaluate the mean change in serum alkaline transaminase from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Aspartate Transaminase Test | 12 weeks
  Evaluate the mean change in aspartate transaminase from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Alkaline Phosphatase Test | 12 weeks
  Evaluate the mean change in Alkaline Phosphatase from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Bilirubin Test | 12 weeks
  Evaluate the mean change in bilirubin from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Serum Creatinine Test | 12 weeks
  Evaluate the mean change in serum creatinine from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Blood Urea Nitrogen Test | 12 weeks
  Evaluate the mean change in blood urea nitrogen from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
T4 | 12 weeks
  Evaluate the mean change in thyroid profile serum thyroxin (T4) from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
T3 | 12 weeks
  Evaluate the mean change in serum triiodothyronine (T3) from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Serum TSH | 12 weeks
  Evaluate the mean change in serum TSH from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
Fasting Blood Sugar | 12 weeks
  Evaluate the mean change in fasting blood sugar from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.
HbA1c | 12 weeks
  Evaluate the mean change in HbA1c from Visit 1 (Screening/Enrollment/Baseline Visit), Visit 2 (Week 4), Visit 3 (Week 8), and Visit 4 (Week 12), end of study in healthy subjects.

SECONDARY OUTCOMES:
Adverse Events | 12 weeks
  Number and proportion of treatment emergent adverse events (TEAEs) and treatment emergent serious adverse event (TESAE) due to Ashwagandha capsules over 12 weeks
Quality of Life (SF-36 QoL) | 12 weeks
  Changes from baseline in the Quality of Life (SF-36 QoL) scores over a period of 12 weeks after start of Ashwagandha

CONTACTS AND LOCATIONS:
Locations (1):
- SF Research Institute, San Francisco, California, United States